## Athens, 15. 11. 2024

ClinicalTrials.gov ID: NCT05623228

Brief Title: The Effectiveness and Efficacy of the Combination of the IntegratedPsychological Therapy and Metacognitive Training. (ATHSCHIZ) (ATH22-24)

Official Title: The Effectiveness and Efficacy of the Combination of the Integrated

Psychological Therapy and Metacognitive Training in Schizophrenia and Treatment Resistant Schizophrenia. This is a Non-randomized Trial. The Therapy Lasts 60 Sessions.

Dr. Stavroula Rakitzi
Clinical psychologist and cognitive behavioral
psychotherapistPrivate practice
ILISION 34
15771 Athens Greece

Tel: +306989766935 srakitzi@gmail.com

Links: URL:

https://www.linkedin.com/

Description linkedin Stavroula

Rakitzi URL: http://orcid.org

Description orcid: 0000-0002-5231-6619

Dr. Polyxeni Georgila
Psychiatrist and cognitive behavioral
psychotherapistPrivate practice
ILISION 34
15771 Athens Greece

15771 Athens Greece Tel: +306932905259

polyxenigeorgila@gmail.com

Links: URL:

https://www.linkedin.com/

Description linkedin Polyxeni

GeorgilaURL: http://orcid.org Orcid:0000-0003-3137-506X

## **Informed Consent to the research protocol**

Dr. Stavroula Rakitzi, a clinical psychologist and cognitive behavioral psychotherapist, and Mrs. Polyxeni Georgila, M.D., psychiatrist, apply a group cognitive behavioral rehabilitation psychotherapy, in which the Integrated Psychological Therapy & Metacognitive Training treatments will be implemented. These treatments aim to improve cognitive functions, symptoms, social and problem-solving skills, as well as restructuring negative thoughts. These groups will start on 28. 11. 2022 and will take place twice a week in one-hour sessions. They will last 60 sessions. Psychological tests will be administered before the start of the treatment, after the intervention and 6 months after the end of the intervention. Up to 5 excused absences are allowed. The goal of these groups is to improve quality of life and rehabilitation. At the same time, the effectiveness of this intervention will be investigated. This means that the test results will be used for statistical analysis to investigate the effectiveness of the treatment. Results will be anonymous, and no personal data will be displayed from any individual participating in the groups. I will let you know about the results. My participation in these groups is voluntary. I certify that I have been informed of the above and that I agree with them.

Athens, Name-surname Signature